CLINICAL TRIAL: NCT05674669
Title: A Phase 1, Single-centre, Dose-escalation Study Utilising Both Open-label and Double-blind Placebo-controlled Crossover Design Studies to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Low Doses of Lysergic Acid Diethylamide Ranging From 50 µg to 100 µg in Healthy Volunteers
Brief Title: A Dose-Ranging Study of 50 µg to 100 µg LSD in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eleusis Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: CAS-50-37-3-02; 2015-003151-21 (EudraCT Number)
Record Dates: First submitted 2022-07-27; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Healthy
MeSH Terms: interventions — Lysergic Acid Diethylamide

STUDY DESIGN:
Intervention Model Description: In Part 1, each subject was allocated to open label treatment with a single dose of 50 µg, 75 µg, or 100 µg LSD. Part 1 was conducted in hallucinogen non-naive participants. In Part 2, each subject was randomized to double blind treatment and received 50 µg LSD followed by 75 µg LSD (experimental non-crossover group), or placebo followed by 75 µg LSD (placebo-controlled crossover group), with dosing separated by at least 7 days. Part 2 was conducted in hallucinogen naive participants.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1 N=3 (Experimental): Single dose, follow-up visits at one day, one week, and one month after dose.
  Interventions: Drug: Lysergic Acid Diethylamide (LSD) 50µg
- Group 2 N=7 (Experimental): Single dose, follow-up visits at one day, one week, and one month after dose.
  Interventions: Drug: Lysergic Acid Diethylamide (LSD) 75µg
- Group 3 N=3 (Experimental): Single dose, follow-up visits at one day, one week, and one month after dose.
  Interventions: Drug: Lysergic Acid Diethylamide (LSD) 100µg
- Group 4 N=10 (Experimental): Randomized treatment with placebo followed by single dose, separated by 7 days. Follow-up visits at one day, one week, and one month after last dose.
  Interventions: Drug: Placebo/Lysergic Acid Diethylamide (LSD) 75µg
- Group 5 N=9 (Experimental): Randomized treatment with single dose followed by second dose, separated by 7 days. Follow-up visits at one day, one week, and one month after last dose.
  Interventions: Drug: Lysergic Acid Diethylamide (LSD) 50µg/75µg

INTERVENTIONS:
Drug: Lysergic Acid Diethylamide (LSD) 50µg
  Arms: Group 1 N=3
Drug: Lysergic Acid Diethylamide (LSD) 75µg
  Arms: Group 2 N=7
Drug: Lysergic Acid Diethylamide (LSD) 100µg
  Arms: Group 3 N=3
Drug: Placebo/Lysergic Acid Diethylamide (LSD) 75µg
  Arms: Group 4 N=10
Drug: Lysergic Acid Diethylamide (LSD) 50µg/75µg
  Arms: Group 5 N=9

SUMMARY:
This study with low-dose LSD comprised 2 substudies in healthy subjects. Subjects who met all inclusion and no exclusion criteria provided written informed consent. Part 1 was an open-label dose-escalation study in hallucinogen non-naïve subjects with significant prior experience with hallucinogens, during which each subject received a single dose of LSD: 50, 75, or 100 µg. Part 2 was a double blind, placebo controlled, randomised, crossover study in hallucinogen naïve subjects with no prior experience with hallucinogens in the last 7 years, during which each subject was assigned to 1 of 8 cohorts and then randomly assigned to receive single doses of LSD 50 µg followed by 75 µg, or placebo followed by 75 µg, with dosing separated by at least 7 days. Subjects were followed up on the day after each dosing, and 1 week and 1 month after the last dose of study treatment. A total of 32 subjects were enrolled.

DETAILED DESCRIPTION:
This study with low-dose LSD comprised 2 substudies in different populations of healthy subjects:

Part 1: an open-label dose-escalation study in hallucinogen non-naïve subjects. Part 2: a double blind, placebo controlled, randomised, crossover study in hallucinogen naïve subjects.

Part 1: Open-label, dose escalation study This part was performed in a population of healthy subjects with significant prior experience with hallucinogens. There was a screening period of up to 28 days. Following provision of informed consent and completion of all screening assessments, eligible subjects were assigned to the open-label dose-escalation group.

Following completion of baseline assessments, each subject received a single dose of LSD: 50, 75, or 100 µg. This dose range was selected for assessment based on extensive historical and clinical LSD research. Subjects knew they would receive the experimental drug but were blinded to the dose level received. Subjects were followed up on the day after dosing and at 1 week and 1 month after dosing.

During screening, baseline, treatment, and follow-up, subjects underwent a series of assessments. Included amongst these assessments were cognitive tasks that were administered at baseline before administration of LSD and subsequently during the study. The open-label study subjects also provided samples for PK analysis.

Part 2: Double-blind, placebo controlled, randomised, crossover study This part commenced following evaluation of the results from Part 1. It was performed in a population of healthy subjects with no prior experience with hallucinogens during the last 7 years. There was a screening period of up to 28 days. Following provision of informed consent and completion of all screening assessments, eligible subjects were assigned to 1 of 8 cohorts and then randomly assigned to 1 of 2 treatment groups. Cognitive assessments were administered at baseline before administration of the first dose and subsequently during the study.

Following completion of baseline assessments, subjects entered a 2 week treatment period: the experimental non-crossover group received 2 sequential escalating single doses of LSD administered at levels determined in Part 1 (50 µg followed by 75 µg, or placebo followed by 75 µg), with dosing separated by at least 7 days; the placebo controlled crossover group received placebo followed at least 7 days later by a single dose of 75 µg LSD, as determined in Part 1. Subjects were followed up on the day after each dosing, 1 week after the second dose, and at 1 month after the last dose of study treatment.

During screening, baseline, treatment and follow-up days, subjects underwent a series of assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subject aged 21 to 65 years inclusive.
2. For Part 1, subject has been previously exposed to LSD or any other classic psychedelic drug, including psilocybin, mescaline, and ayahuasca, on more than 3 occasions during their lifetime. For Part 2, Subject has not been previously exposed to LSD or any other classic psychedelic drug, including psilocybin, mescaline, and ayahuasca, during the past 7 years.
3. Subject was able and willing to give written informed consent, adhere to the compliance terms during participation in the study, undergo the examinations and testing set forth in the clinical study protocol, and clearly and reliably communicate their subjective experiences to the investigator.
4. Female participants of childbearing potential and male participants whose partner was of childbearing potential must have been willing to ensure that they or their partner used effective contraception during the study and for 3 months after the final study drug administration.

Exclusion Criteria:

A. General Health

1. Subject had a presence or clinically relevant history of any psychiatric, respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders, as judged by the investigator.
2. Subject had a resting blood pressure exceeding 140 mmHg (systolic) or 90 mmHg (diastolic), averaged across 4 assessments taken at least 1 minute apart on the same day.
3. Subject had a presence or relevant history of organic brain disorders (e.g., intracranial hypertension, aneurisms, impaired consciousness, lethargy, or brain tumour).
4. Subject had a relevant history of atopy, hypersensitivity, skin allergies, or allergic reactions to drugs.
5. Subject had a clinical laboratory test result outside the reference ranges of the testing laboratory and considered clinically significant by the investigator.
6. Subject was positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or human immunodeficiency (HIV) virus I or II at screening.
7. Subject was a current smoker (i.e., had smoked within 1 month prior to the screening visit).
8. Subject had a medical history that would affect the subject's safety or the study endpoints.
9. Subject had used prescription drugs which might potentially interact with the pharmacokinetics of LSD or therapy within 14 days of first dosing, unless agreed as not clinically relevant by the PI and the Medical Monitor.
10. Subject had used over the counter (OTC) medication or therapy, including megadose vitamin therapy (but excluding routine vitamins) within 7 days of first dosing, unless agreed as not clinically relevant by the PI and the Medical Monitor.
11. Subject had donated or received any blood or blood products within the previous 3 months prior to first dosing.
12. Subject could not use a computer to complete simple tasks such as responding to an email.
13. Subject had used any investigational drug or participated in any clinical trial within 3 months of their first dosing.
14. Subject had a current sleep disorder.
15. Subject had a history of cataracts, active glaucoma or any other ophthalmic condition that could interfere with the eye blink assessment.
16. Subject had veins unsuitable for venepuncture and/or cannulation.
17. Subject had a corrected QT interval using Fridericia's correction >450 milliseconds.
18. Subject was unlikely to cooperate with the requirements of the study, in the opinion of the PI or designee.
19. Subject was pregnant or lactating
20. Exclusion Part 2 only: Subject had a history of drug abuse or dependence in the last 12 months, had current drug abuse or dependence or had a positive result for drugs of abuse and alcohol tests at screening or admission.

    B. Psychiatric Health
21. Subject had a current or past history of meeting Diagnostic and Statistical Manual of Mental Disorders fourth edition criteria for schizophrenia or other psychotic disorders (unless substance induced or due to a medical condition), bipolar I or II disorder, a major depressive episode, a manic or hypomanic episode, alcohol dependence or abuse (in the past 5 years), substance dependence and abuse (in the past 5 years), current panic disorder, obsessive compulsive disorder, social anxiety disorder, generalised anxiety disorder, anorexia, bulimia or post-traumatic stress disorder
22. Subject had a first- or second-degree relative with schizophrenia, other psychotic disorders (unless substance-induced or due to a medical condition), or bipolar I or II disorder.
23. Subject was receiving chronic administration of tricyclic antidepressants or lithium or acute administration of serotonin reuptake inhibitors, haloperidol, serotonin reuptake inhibitors or monoamine oxidase inhibitors.
24. Subject was taking OTC doses of 5-hydroxytryptophan or St John's Wort or ayahuasca (which contains monoamine oxidase inhibitors in addition to dimethyltryptamine).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2016-07-26 (Actual); Study Completion 2017-07-17 (Actual)

PRIMARY OUTCOMES:
Assessment of Adverse Events by % frequency | 1 year
  Assessment of Adverse Events by % frequency to assess the safety and tolerability of LSD
AUC 0-24h ( pg/mL*h) over time | 24 hours
  AUC 0-24h ( pg/mL*h): area under the plasma concentration-time curve profiles from time zero to the 24 hour sample determined using the linear trapezoidal rule
Cmax (pg/mL)drug | 24 hours
  Cmax (pg/mL): maximum drug plasma concentration
Tmax (h) | 24 hours
  Tmax (h): time to reach maximum plasma concentration, T1/2 (h): time to reach half of maximum drug plasma concentration

SECONDARY OUTCOMES:
Assess subjective drug effects using a VAS. | 12 hours
  Assessed by the Visual Analog Scale (VAS). Items assess acute subjective drug effects (e.g. intensity, liking) Item scores are assessed on a visual scale ranging from 1% to 100%. Higher scores indicate greater subjective effects
Assess subjective drug effects on the 5D-ASC | 12 hours
  5-Dimensional Altered States of Consciousness Questionnaire (5D-ASC). The scale ranges from no, not more than usual (on the left) to yes, very much more than usual (on the right). Items retrospectively assess subjective drug effects. Item scores are assessed on a visual scale ranging from 1% to 100%. Higher scores indicate greater subjective effects associated with a different state of consciousness
Assess ego dissolution by the EDI | 12 hours
  The EDI is an eight-item questionnaire designed to measure ego dissolution. Each item is scored on a 5-point Likert-type scale, and the inventory includes a single factor. Higher scores indicate greater subjective effects associated with a different state of consciousness
Assess the characteristics of altered states of consciousness assessed by the MEQ | 12 hours
  The MEQ is a 30-item self-report questionnaire developed for detecting and characterizing mystical experiences induced by classic psychedelics. Each item is scored on a 5-point Likert-type scale, and derived scores for the MEQ include four scales: mystical, positive mood, transcendence of time and space, and ineffability. In addition, a response of more than or equal to 60% of each and every scale would classify an experience as a 'complete mystical experience'. Higher scores indicate greater subjective effects associated with a different state of consciousness.

CONTACTS AND LOCATIONS:
Overall Officials: Director of Research and Development, Study Director — Eleusis Therapeutics
Locations (1):
- PAREXEL, Early Phase Clinical Unit, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No